CLINICAL TRIAL: NCT02029365
Title: Single-center Study, Transversal, Controlled and Not Randomized, Laying on the Desire of Children and Eating Disorders in a Population of Infertile Women
Brief Title: Transversal, Controlled and Not Randomized Study, Laying on the Desire of Children and Eating Disorders in a Population of Infertile Women
Acronym: TCA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC13_0449
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Infertility; Eating Disorders
Keywords: Infertility; desire for children; eating disorder; anorexia nervosa; bulimia nervosa; eating disorders not otherwise specified
MeSH Terms: conditions — Infertility; Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Without eating disorders (Other): Women consulting for infertility but without diagnosis of eating disorder.
  Interventions: Other: Autoquestionnary
- With Eating disorders (Other): Womenconsulting for infertility for which eating disorder is diagnosed.
  Interventions: Other: Autoquestionnary; Other: semi-structured interview

INTERVENTIONS:
Other: Autoquestionnary — autoquestionnary completed during the consultation for infertility
Other: semi-structured interview — phone interview
  Arms: With Eating disorders

SUMMARY:
In France , 15% of couples seek help for problems conceiving . In 10% of cases, infertility remains " unexplained" . Among the causes of female infertility , there are the eating disorders, as well as sexual disorders , these two cases may be linked. In addition, data from the literature seem to suggest that beyond a diagnosis of eating disorders, the feeding behavior of infertile women is more often disturbed than the general population. Moreover, the notions of desire for a child and maternal representations seem essential to address in the comprehensive care of women with infertility but also TCA integrating all conflicting issues reactivated at the time of motherhood. However, little work has been done on this subject. Thus, we propose a study on the desire for children and the eating disorders to infertile women, to update epidemiological data, but also to better characterize this particular patient population. Perspectives of this work are to improve screening measures and support through a joint work of doctors reproductive and psychiatrists.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Major
* In a relationship
* Infertile (WHO criteria)
* Consultant in the Department of infertility (BMDR) for AMP
* Understanding of French, literate
* Agree to participate in the study

Exclusion Criteria:

* Man
* Minor
* Pregnancy at the time of assessment
* Exclusive Infertility spouse
* Disorders of higher functions (severe cognitive impairment or confusion) or psychosis (hallucinations, delusional syndrome)
* Major protected

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Children desire | 30 days
  Questionnaire scores of children desire (Fragebogen zum Kinderwunsch) , according to three dimensions:
  * Improved self-esteem''
  * Emotional Stabilization
  * Ambivalence

SECONDARY OUTCOMES:
Dysmorphic | 30 days
  score Body Shape Questionnaire (BSQ)
Sexuality | 30 days
  History Questionnaire score Sexual (QHS)
Anxiety and depression | 30 days
  score on the Hospital Anxiety and Depression Scale (HAD)
Quality of life questionnaire | 30 days
  Quality of life questionnaire score FertiQol internationnal

CONTACTS AND LOCATIONS:
Overall Officials: Marie GRALL-BRONNEC, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes university Hospital, Nantes, France